CLINICAL TRIAL: NCT05584046
Title: Effect of a Novel Herbal Patch for the Treatment of Plantar Fasciitis - A Single-blind Randomized Controlled Trial
Brief Title: A Single-blind RCT to Investigate the Effect of a Novel Herbal Patch for the Treatment of PF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Pauline Lui, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.426
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Plantar Fasciitis
Keywords: Plantar Fasciitis; Herbal Patch
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDAM group (Experimental): Patients receive the CDAM patch and a standard home stretching exercise program
  Interventions: Other: CDAM
- Untreated group (No Intervention): Patients receive a standard home stretching exercise program

INTERVENTIONS:
Other: CDAM — Novel drugs such as Traditional Chinese Medicine (TCM) formula that can suppress inflammation may augment tissue healing and reduce activity-related pain in patients suffering from plantar fasciitis. Our team has experiences of using TCM for the treatment of plantar fasciitis. Based on our previous experience, our group has developed a new proprietary topical TCM herbal formula, CDAM, containing Carthami Flos , Dipsaci Radix , Aconiti Lateralis Radix Praeparata and Herba Menthae for the treatment of plantar fasciitis.
  Arms: CDAM group

SUMMARY:
Disorders and injuries of tendons and ligaments are some of the most diagnosed musculoskeletal (MS) disorders clinically. Nearly half of the 33 million MS disorders reported in the United States each year are tendon and ligament injuries. Although most of such injuries are non-fatal, they are severely debilitating, resulting in significant reduction in patient's quality of life, loss of productivity, and considerable costs to the healthcare system.

Among all tendon and ligament disorders and injuries, tendon and ligament overuse disorders are the most common and incapacitating ones. Tendinopathy is a painful tendon overuse disorder, which increases with population aging. It has been estimated that about 30% of consultations for MS complaints in a general practice were related to tendinopathy. The affected tendon is presented with local tenderness, swelling and pain, causing physical disability of the affected individual. The affected tendon degenerates and finally ruptures. Common sites of tendinopathy include supraspinatus, common wrist extensor, flexor tendon, patellar tendon, and Achilles tendon. The outcomes of both conservative treatments and surgeries are not satisfactory, with recurrent pain and tendon retear after surgery.

Plantar fasciitis is a chronic painful, degenerative condition of the plantar fascia. It is caused by repetitive traumas at its origin on the calcaneus. Plantar fascia is a thick, ribbon-like fibrous ligament that connects the medial calcaneal tubercle to the heads of the metatarsal bones. It contributes to the support of the foot arch by acting as a tie-rod, where it undergoes tension when the foot bears weight. Therefore, although plantar fascia is anatomically defined as a ligament, it functions similar to a tendon.

This study aims to conduct a randomized controlled study to test the efficacy of CDAM patch for the treatment of plantar fasciitis in patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female with age 18-65
* Unilateral or bilateral
* Heel pain for more than 6 weeks' duration
* VAS score ≥ 5
* Signed informed consent.

Exclusion Criteria:

* Known chronic disease or receiving long-term medications affecting bone metabolism including BPs
* Contraindication to alendronate therapy such as poor dental fitness
* ACL injury less than 6 weeks
* Injury on duty cases
* Patients who have undergone arthroscopy or open surgery in the index knee in the last 12 months
* Other associated injuries (fractures and other ligament involvement such as neurovascular bundles injury)
* Chondral lesion with concomitant intervention
* Presence of X-ray features of osteoarthritis including decrease in joint space, presence of osteophytes and subchondral cysts
* Neurological deficit
* Pregnant or breastfeeding
* Inability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Foot Function Index (FFI) questionnaire | Change from baseline FFI at 3 weeks
  The FFI consists of 23 self-reported items divided into three subscales: limitation, pain and disability. The items are scored on a 10-point Likert scale. For each subscale, the raw score is transformed to a 100-point score, with higher score indicating worse limitation / pain / disability. The total score of FFI is the mean of the subscale scores. The Taiwan Chinese version of FFI has been validated.
Foot Function Index (FFI) questionnaire | Change from baseline FFI at 6 weeks
  The FFI consists of 23 self-reported items divided into three subscales: limitation, pain and disability. The items are scored on a 10-point Likert scale. For each subscale, the raw score is transformed to a 100-point score, with higher score indicating worse limitation / pain / disability. The total score of FFI is the mean of the subscale scores. The Taiwan Chinese version of FFI has been validated.
Foot Function Index (FFI) questionnaire | Change from baseline FFI at 8 weeks
  The FFI consists of 23 self-reported items divided into three subscales: limitation, pain and disability. The items are scored on a 10-point Likert scale. For each subscale, the raw score is transformed to a 100-point score, with higher score indicating worse limitation / pain / disability. The total score of FFI is the mean of the subscale scores. The Taiwan Chinese version of FFI has been validated.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong